CLINICAL TRIAL: NCT00092014
Title: A 12-Month Extension to: A Randomized, Double-Blind, Double-Dummy, Parallel-Group, Multicenter Study to Evaluate and Compare the Effects of Once Weekly Alendronate and Risedronate on Bone Mineral Density in Postmenopausal Women With Osteoporosis
Brief Title: A Study to Evaluate and Compare Alendronate and Risedronate on Bone Mineral Density in Women With Postmenopausal Osteoporosis (MK-0217-211)
Acronym: FACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217-211; 2004_016 (Other: Protocol number)
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2024-04

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate; Risedronic Acid; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alendronate 70 mg (Experimental): Alendronate sodium, 70 mg, orally once weekly for up to 24 months
  Interventions: Drug: Alendronate; Dietary Supplement: Elemental Calcium; Dietary Supplement: Vitamin D; Drug: Risendronate placebo
- Risendronate 35 mg (Active Comparator): Risendronate, 35 mg, orally once weekly for up to 24 months
  Interventions: Drug: Risedronate 35 mg; Dietary Supplement: Elemental Calcium; Dietary Supplement: Vitamin D; Drug: Alendronate placebo

INTERVENTIONS:
Drug: Alendronate — Alendronate sodium, 70 mg, once weekly for up to 24 months. Medications were taken fasting which was maintained for 30 minutes postdose.
  Other Names: MK-0217; FOSAMAX®
  Arms: Alendronate 70 mg
Drug: Risedronate 35 mg — Risendronate, 35 mg, once weekly for up to 24 months. Medications were taken fasting which was maintained for 30 minutes postdose.
  Other Names: Actonel®; Atelvia®
  Arms: Risendronate 35 mg
Dietary Supplement: Elemental Calcium — Elemental calcium at least 1,000 mg daily (diet plus supplements). Medications were taken fasting which was maintained for 30 minutes postdose.
Dietary Supplement: Vitamin D — Vitamin D at least 400 international units daily (diet plus supplements). Medications were taken fasting which was maintained for 30 minutes postdose.
Drug: Risendronate placebo — Risendronate placebo was taken once weekly for up to 24 months. Medications were taken fasting which was maintained for 30 minutes postdose.
  Arms: Alendronate 70 mg
Drug: Alendronate placebo — Alendronate placebo was taken once weekly for up to 24 months. Medications were taken fasting which was maintained for 30 minutes postdose.
  Arms: Risendronate 35 mg

SUMMARY:
This study is to evaluate and compare the effects of Alendronate and Risedronate to treat women with postmenopausal osteoporosis. The primary hypothesis for this study is that in postmenopausal women with osteoporosis, treatment with oral alendronate 70 mg once weekly will produce a mean percent increase from baseline in hip trochanter bone mineral density (BMD) at 12 and 24 months which is greater than that observed with oral risedronate 35 mg once weekly.

ELIGIBILITY:
Inclusion Criteria:

* Women with postmenopausal osteoporosis

Exclusion Criteria:

* Bilateral hip replacements
* Esophageal abnormalities
* Metabolic bone disease (example - Vitamin D deficiency)
* Medications that would affect the breakdown or build-up of bone turnover

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2002-09-01 (Actual); Primary Completion 2004-04-01 (Actual); Study Completion 2004-04-01 (Actual)

PRIMARY OUTCOMES:
Mean percent change from baseline in hip trochanter bone mineral density (BMD) at 12 months | Baseline and 12 months
Mean percent change from baseline in hip trochanter BMD at 24 months | Baseline and 24 months

SECONDARY OUTCOMES:
Mean percent change from baseline in total hip, femoral neck, posteroanterior (PA) lumbar BMD at 12 months | Baseline and 12 months
Mean percent change from baseline in total hip, femoral neck, posteroanterior (PA) lumbar BMD at 24 months | Baseline and 24 months
Change from baseline in biochemical markers of bone turnover at 12 months | Baseline and 12 months
Change from baseline in biochemical markers of bone turnover at 24 months | Baseline and 24 months
Percent responders (>=0% and >=3% change from baseline in hip trochanter and lumbar spine BMD) at 12 months | 12 months
Percent responders ((>=0% and >=3% change from baseline in hip trochanter and lumbar spine BMD) at 24 months | 24 months
Number of participants who experienced one or more adverse events (AE) | Up to 24 months
Number of participants who discontinued study medication due to an AE | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Rosen CJ, Hochberg MC, Bonnick SL, McClung M, Miller P, Broy S, Kagan R, Chen E, Petruschke RA, Thompson DE, de Papp AE; Fosamax Actonel Comparison Trial Investigators. Treatment with once-weekly alendronate 70 mg compared with once-weekly risedronate 35 mg in women with postmenopausal osteoporosis: a randomized double-blind study. J Bone Miner Res. 2005 Jan;20(1):141-51. doi: 10.1359/JBMR.040920. Epub 2004 Sep 29. PMID 15619680
- [Background] Sebba AI, Bonnick SL, Kagan R, Thompson DE, Skalky CS, Chen E, de Papp AE; Fosamax Actonel Comparison Trial investigators. Response to therapy with once-weekly alendronate 70 mg compared to once-weekly risedronate 35 mg in the treatment of postmenopausal osteoporosis. Curr Med Res Opin. 2004 Dec;20(12):2031-41. doi: 10.1185/030079904x16768. PMID 15706659
- [Background] Bonnick S, Saag KG, Kiel DP, McClung M, Hochberg M, Burnett SM, Sebba A, Kagan R, Chen E, Thompson DE, de Papp AE. Comparison of weekly treatment of postmenopausal osteoporosis with alendronate versus risedronate over two years. J Clin Endocrinol Metab. 2006 Jul;91(7):2631-7. doi: 10.1210/jc.2005-2602. Epub 2006 Apr 24. PMID 16636120
- [Background] Burnett-Bowie SM, Saag K, Sebba A, de Papp AE, Chen E, Rosenberg E, Greenspan SL. Prediction of changes in bone mineral density in postmenopausal women treated with once-weekly bisphosphonates. J Clin Endocrinol Metab. 2009 Apr;94(4):1097-103. doi: 10.1210/jc.2008-1122. Epub 2009 Jan 13. PMID 19141590